CLINICAL TRIAL: NCT02724579
Title: A Phase 2 Study of Reduced Therapy for Newly Diagnosed Average-Risk WNT-Driven Medulloblastoma Patients
Brief Title: Reduced Craniospinal Radiation Therapy and Chemotherapy in Treating Younger Patients With Newly Diagnosed WNT-Driven Medulloblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACNS1422; NCI-2016-00150 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACNS1422 (Other: Children's Oncology Group); ACNS1422 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2016-03-25; First posted 2016-03-31 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-02

CONDITIONS: Medulloblastoma
MeSH Terms: conditions — Medulloblastoma | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cyclophosphamide; Lomustine; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (reduced radiation therapy and chemotherapy) (Experimental): RADIATION THERAPY: Beginning 4-5 weeks after surgery, patients undergo craniospinal radiation therapy 5 days a week for 6 weeks.
  MAINTENANCE THERAPY (WEEKS 1, 3, 5, and 7): Beginning 4-6 weeks after completion of radiation therapy patients receive lomustine PO on day 1, vincristine sulfate IV over 1 minute or via minibag on days 1, 8, and 15, and cisplatin IV over 6 hours on day 1. Treatment repeats every 42 days in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY (WEEKS 2, 4, AND 6): Patients receive cyclophosphamide IV over 30-60 minutes on days 1 and 2, mesna IV over 15-30 minutes on days 1 and 2, and vincristine sulfate IV over 1 minute or via minibag on days 1 and 8. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Patients also undergo MRI throughout the trial.
  Interventions: Drug: Cisplatin; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Drug: Lomustine; Procedure: Magnetic Resonance Imaging; Radiation: Radiation Therapy; Drug: Vincristine; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lomustine — Given PO
  Other Names: 1-(2-Chloroethyl)-3-cyclohexyl-1-nitrosourea; 1-Nitrosourea, 1-(2-chloroethyl)-3-cyclohexyl-; Belustin; Belustine; CCNU; Cecenu; CeeNU; Chloroethylcyclohexylnitrosourea; Citostal; Gleostine; Lomeblastin; Lomustinum; Lucostin; Lucostine; N-(2-Chloroethyl)-N'-cyclohexyl-N-nitrosourea; Prava; RB-1509; WR-139017
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Radiation: Radiation Therapy — Undergo craniospinal radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Vincristine — Given IV or via minibag
  Other Names: LCR; Leurocristine; VCR; Vincrystine
Drug: Vincristine Sulfate — Given IV or via minibag
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies how well reduced doses of radiation therapy to the brain and spine (craniospinal) and chemotherapy work in treating patients with newly diagnosed type of brain tumor called WNT)/Wingless (WNT)-driven medulloblastoma. Recent studies using chemotherapy and radiation therapy have been shown to be effective in treating patients with WNT-driven medulloblastoma. However, there is a concern about the late side effects of treatment, such as learning difficulties, lower amounts of hormones, or other problems in performing daily activities. Radiotherapy uses high-energy radiation from x-rays to kill cancer cells and shrink tumors. Drugs used in chemotherapy, such as cisplatin, vincristine sulfate, cyclophosphamide and lomustine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving reduced craniospinal radiation therapy and chemotherapy may kill tumor cells and may also reduce the late side effects of treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the progression-free survival (PFS) of children >= 3 years of age with wingless-type MMTV integration site family (WNT)-driven average-risk medulloblastoma using reduced craniospinal radiotherapy (CSI) (18 Gray [Gy]) with a limited target volume boost to the tumor bed of 36 Gy for a total of 54 Gy and reduced chemotherapy approach (no vincristine [vincristine sulfate] during radiotherapy and reduced-dose maintenance chemotherapy) and to monitor the PFS for early evidence that the outcome is unacceptable.

SECONDARY OBJECTIVES:

I. To prospectively test the hypothesis that deoxyribonucleic acid (DNA) methylation profiling will accurately classify WNT-driven medulloblastoma.

II. To prospectively evaluate and longitudinally model the cognitive, social, emotional, behavioral, and quality of life (QoL) functioning of children who are treated with reduced CSI (18 Gy) with a limited target volume boost to the tumor bed (to a total of 54 Gy) and reduced chemotherapy (reduced cisplatin, vincristine, and lomustine [CCNU]).

EXPLORATORY OBJECTIVES:

I. To explore whether DNA methylation profiling of medulloblastoma samples will result in a predictive classification scheme for the Sonic Hedgehog (SHH), Group 3, and Group 4 medulloblastoma subgroups according to the Heidelberg classifier. This will be addressed in a separate biology protocol.

II. To describe the audiologic and endocrinologic toxicities, as well as peripheral neuropathy, in children treated with reduced CSI (18 Gy) with a limited target volume boost to the tumor bed (to a total of 54 Gy) and reduced cisplatin and vincristine chemotherapy.

OUTLINE:

RADIATION THERAPY: Beginning 4-5 weeks after surgery, patients undergo craniospinal radiation therapy 5 days a week for 6 weeks.

MAINTENANCE THERAPY (WEEKS 1, 3, 5, and 7): Beginning 4-6 weeks after completion of radiation therapy patients receive lomustine orally (PO) on day 1, vincristine sulfate intravenously (IV) via minibag on days 1, 8, and 15, and cisplatin IV over 6 hours on day 1. Treatment repeats every 42 days in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY (WEEKS 2, 4, AND 6): Patients receive cyclophosphamide IV over 30-60 minutes on days 1 and 2, mesna IV over 15-30 minutes on days 1 and 2, and vincristine sulfate IV via minibag on days 1 and 8. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients also undergo magnetic resonance imaging (MRI) throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 2 years, and then annually for 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be greater than or equal to 3 years and less than 22 years of age at the time of enrollment
* Patients must be newly diagnosed and have:

  * Eligibility confirmed by rapid central pathology and molecular screening review on APEC14B1:

    * Classical histologic type (non LC/A) WNT medulloblastoma
    * Positive nuclear beta-catenin by immunohistochemistry (IHC)
    * Positive for CTNNB1 mutation by Sanger sequencing
    * Negative for MYC and MYCN by fluorescence in situ hybridization (FISH)
* Patient must have negative lumbar cerebrospinal fluid (CSF) cytology

  * Note: CSF cytology for staging should be performed no sooner than 14 days post operatively to avoid false positive CSF; ideally, CSF should be obtained between day 14 and day 21 to allow for final staging status before enrollment onto the study; patients with positive CSF cytology obtained 0 to 14 days after surgery should have cytology repeated to determine eligibility and final CSF status; patients with negative CSF cytology from lumbar puncture obtained 0 to 14 days after surgery do not need cytology repeated; patients with negative CSF cytology from lumbar puncture obtained prior to surgery do not need cytology repeated post-operatively
* Patients must have eligibility confirmed by Rapid Central Imaging Review on APEC14B1; patients must have =< 1.5 cm^2 maximal cross-sectional area of residual tumor; whole brain magnetic resonance imaging (MRI) with and without gadolinium and spine MRI with gadolinium must be performed
* Patients must be enrolled, and protocol therapy must be projected to begin, no later than 36 days after definitive diagnostic surgery (day 0)
* Peripheral absolute neutrophil count (ANC) >= 1000/uL
* Platelet count >= 100,000/uL (transfusion independent)
* Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 3 to < 6 years of age: maximum (max) serum creatinine 0.8 mg/dL (males and females)
  * 6 to < 10 years of age: max serum creatinine 1 mg/dL (males and females)
  * 10 to < 13 years of age: max serum creatinine 1.2 mg/dL (males and females)
  * 13 to < 16 years of age: max serum creatinine 1.5 md/dL (males) and 1.4 md/dL (females)
  * >= 16 years of age: max serum creatinine 1.7 mg/dL (males) and 1.4 mg/dL (females)

    * The threshold creatinine values were derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the Centers for Disease Control and Prevention (CDC)
* Total or direct bilirubin =< 1.5 x upper limit of normal (ULN) for age, and
* Serum glutamate pyruvate (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L (3x ULN); for the purpose of this study, the ULN for SGPT is 45 U/L
* Central nervous system function defined as:

  * Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled
  * Patients must not be in status epilepticus, a coma or on assisted ventilation at the time of study enrollment
* Patients must have receptive and expressive language skills in English, French, or Spanish to complete the QoL and neurocognitive assessments; if a patient meets these criteria but the parent/guardian speaks a language other than English, French, or Spanish, the patient may still be enrolled and tested, and the parent-report measures should be omitted
* All patients and/or their parents or legal guardians must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with metastatic disease by either MRI evaluation (brain and spine) or lumbar CSF cytology are not eligible; patients who are unable to undergo a lumbar puncture for assessment of CSF cytology are ineligible
* Patients must not have received any prior radiation therapy or chemotherapy (tumor-directed therapy) other than surgical intervention and/or corticosteroids
* Pregnancy and Breast Feeding

  * Female patients who are pregnant are ineligible due to risks of fetal and teratogenic adverse events as seen in animal/human studies
  * Lactating females are not eligible unless they have agreed not to breastfeed their infants
  * Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained
  * Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation
* Patients with a history of moderate to profound intellectual disability (i.e., intelligence quotient [Q)]=< 55) are not eligible for enrollment; PLEASE NOTE: Children with a prior history of attention deficit hyperactivity disorder (ADHD) or a specific learning disability (e.g., dyslexia) are eligible for this study. Children with posterior fossa syndrome (also known as cerebellar mutism) are eligible for this study

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-11-17 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From the initiation of protocol treatment to the occurrence of any of the following events: disease progression or disease recurrence or death from any cause, assessed up to 10 years
  PFS along with the confidence intervals will be estimated using the Kaplan-Meier method. PFS will also be reported based on central radiology review.

SECONDARY OUTCOMES:
Deoxyribonucleic acid (DNA) methylation profiling as real-time classification of WNT-driven medulloblastoma | Within 32 days of definitive surgery
  Results will be compared to the results of the molecular screening tests. The sensitivity and specificity comparison between DNA methylation arrays and the standard methods (molecular screening tests for WNT using immunohistochemistry [IHC] and CTNNB1 sequencing) will be performed using McNemar's test.
Change in neurocognitive function (cognitive, social, emotional and behavioral) according to Children Oncology Group Standard Neuropsychological Battery | Baseline to up to 60 months post-diagnosis
  Neurocognitive function will be measured at 9, 30 and 60 months post diagnosis and will be compared with the neurocognitive outcomes from an age and gender matched ACNS0331 cohort to the WNT patients treated on ACNS1422. Data for all assessments will be available as standardized t-scores. The change over time for each component of the neuropsychological testing will be estimated using the Generalized Estimating Equation (GEE) approach, with the standardized t-scores as the dependent variable and the assessment times as a covariate. Within the ACNS1422 cohort GEE models will also be used to explore associations of changes over time with factors such as gender, age at initiation of radiation therapy, tumor location, number of surgical interventions, etc.

OTHER OUTCOMES:
DNA methylation profiling of medulloblastoma real-time" predictive classification scheme for the SHH, group 3 and group 4 medulloblastoma subgroups according to the Heidelberg classifier | Within 32 days of definitive surgery
  The proportion of patients classified into each medulloblastoma subgroup will be reported.
Audiologic and endocrinologic toxicities | Up to 10 years
  The proportions of children who experienced audiologic, endocrinologic, and peripheral neuropathy toxicities per grade will be estimated along with 95% confidence interval based on an exact binomial distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Gottardo, Principal Investigator — Children's Oncology Group
Locations (195):
- United States (173):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Puerto Rico (2):
  - HIMA San Pablo Oncologic Hospital, Caguas
  - University Pediatric Hospital, San Juan
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia